CLINICAL TRIAL: NCT01375270
Title: The Effects of Experimental Elevation of Plasma Glucose and Lipid on Pancreatic Beta-cell Function in Humans
Brief Title: Glucolipotoxicity and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Group Leader, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-3-2010-127
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; incretin; beta-cell function; glucolipotoxicity; glucagon-like peptide 1; glucose-dependent insulinotropic polypeptide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucotoxicity Trial (Experimental): Insulin secretion will be assessed using a hyperglycemic clamp combined with GLP-1, GIP, and arginine infusions.
  The clamp will be performed before and after 24 hours of bed rest, isocaloric meal feeding, and experimental elevation of blood glucose.
  Interventions: Procedure: Glucotoxicity
- Control Trial (No Intervention): Insulin secretion will be assessed using a hyperglycemic clamp combined with GLP-1, GIP, and arginine infusions.
  The clamp will be performed before and after 24 hours of bed rest and isocaloric meal feeding.
- Lipotoxicity Trial (Experimental): Insulin secretion will be assessed using a hyperglycemic clamp combined with GLP-1, GIP, and arginine infusions.
  The clamp will be performed before and after 24 hours of bed rest, isocaloric meal feeding, and experimental elevation of blood free fatty acids.
  Interventions: Procedure: Lipotoxicity

INTERVENTIONS:
Procedure: Glucotoxicity — Glucose will be infused intravenously for a 24 hour period to raise blood glucose concentrations 5 mM above basal.
  Arms: Glucotoxicity Trial
Procedure: Lipotoxicity — Intralipid and heparin will be infused intravenously for a 24 hour period to raise blood free fatty acid concentrations to approximately 1 mM.
  Arms: Lipotoxicity Trial

SUMMARY:
Elevations of blood glucose and lipid are thought to be deleterious to the insulin secretory function of the pancreas. This is known as glucolipotoxicity. However, few studies have examined this in detail. This investigation will examine pancreatic insulin secretory function in physiological models of glucolipotoxicity such as obese and type 2 diabetic individuals. Furthermore, healthy subjects will undergo 24 hour infusion of glucose or Intralipid to induce experimental models of glucolipotoxicity. Insulin secretion in response to intravenous infusions of glucose, GLP-1, GIP, and arginine and in response to meal ingestion, will be examined. the investigators hypothesize that experimental glucolipotoxicity will impairs pancreatic insulin secretory function to levels akin to that seen in type 2 diabetics.

ELIGIBILITY:
Inclusion Criteria:

* normal glucose tolerance based on screening OGTT or
* diagnosed type 2 diabetic (confirmed with OGTT)

Exclusion Criteria:

* insulin dependent diabetes
* age <18 or >65 years
* BMI <20 or > 35 kg/m2
* evidence of hematological, pulmonary, hepatic, renal, or cardiovascular disease
* actively undergoing weight-loss (>2kg change in last 6 months)
* bariatric surgery (gastric by-pass or banding)
* pregnancy
* smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Insulin Secretion | 24 hours
  Insulin secretion will be assessed in response to intravenous infusions of glucose, GLP-1, GIP, and arginine, and in response to meal ingestion.

SECONDARY OUTCOMES:
Insulin Sensitivity | 24 hours
  Glucose kinetics will be assesed using [6,6-2H2]glucose. Rate of glucose disappearance during glucose infusion will be quantified per unit of plasma insulin to derive an estimate of insulin sensitivity.
Plasma Cytokines (IL-6, TNF, IL-1beta, IL-1ra) | 24 hours
  Cytokines will be measured in plasma: IL-6, TNF-alpha, IL-1beta, IL-1 receptor antagonist, IL-8, IL-10, Interferon gamma. Peripheral blood mononuclear cells will be isolated.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Solomon, Ph.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Centre of Inflammation and Metabolism, Rigshospitalet, Copenhagen, Denmark